CLINICAL TRIAL: NCT07207668
Title: Effectiveness of Injectable Platelet Rich Fibrin Used For Root Surface Biomodification On Clinical Periodontal Parameters
Brief Title: i-PRF & Root Surface Biomodification
Acronym: iPRF-Perio
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Halil Ata BIÇAKÇIOGLU (Other)
Responsible Party: Sponsor-Investigator, Halil Ata BIÇAKÇIOGLU, Principal Investigator, PhD, Department of Periodontology, Gazi University Faculty of Dentistry, Gazi University
Organization: Gazi University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GÜDHKAEK.2022.24/2; GÜDHKAEK.2022.24/2 (Registry Identifier: Gazi University Faculty of Dentistry Clinical Research Ethics Committee)
Record Dates: First submitted 2025-09-18; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Chronic Periodontitis (Disorder); Periodontitis
Keywords: Open Flap Debridement (OFD); Pro-angiogenic agents; Growth differentiation factors; Immunomodulation; Ethylenediaminetetraacetic Acid (EDTA); Periodontitis; Periodontal Pocket; Root Surface Conditioning; Platelet-Rich Fibrin; Autologous Blood Transfusion
MeSH Terms: conditions — Chronic Periodontitis; Periodontitis; Periodontal Pocket | interventions — proliferation regulatory factors, human urine

STUDY DESIGN:
Intervention Model Description: This is a single-center, randomized, parallel-group trial. Both groups received open flap debridement with 24% EDTA root surface conditioning. In the test group, injectable platelet-rich fibrin (i-PRF) was additionally applied to the surgical sites, whereas in the control group no i-PRF was used. The only difference between groups was the adjunctive use of i-PRF.
Who Masked: Participant
Masking Description: Participants were blinded to group allocation; however, investigators and outcome assessors were not blinded due to the surgical nature of the interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control - OFD + EDTA (Active Comparator): Participants received open flap debridement (OFD) with 24% EDTA root surface conditioning only. No injectable platelet-rich fibrin (i-PRF) was applied.
  Interventions: Procedure: Open Flap Debridement (OFD); Other: 24% EDTA Root Conditioning
- Test - OFD + EDTA + i-PRF (Experimental): Participants received open flap debridement (OFD) with 24% EDTA root surface conditioning plus application of injectable platelet-rich fibrin (i-PRF) to the surgical sites before flap closure.
  Interventions: Procedure: Open Flap Debridement (OFD); Other: 24% EDTA Root Conditioning; Biological: Injectable Platelet-Rich Fibrin (i-PRF)

INTERVENTIONS:
Procedure: Open Flap Debridement (OFD) — Standard periodontal surgical procedure involving full-thickness flap elevation, scaling, and root planing to eliminate inflamed tissue and reduce periodontal pocket depth.
  Other Names: Periodontal Flap Surgery
Other: 24% EDTA Root Conditioning — Application of 24% neutral pH EDTA gel for 3 minutes on root surfaces to remove the smear layer and expose collagen fibers before closure.
  Other Names: Ethylenediaminetetraacetic Acid Gel
Biological: Injectable Platelet-Rich Fibrin (i-PRF) — Autologous platelet concentrate prepared by low-speed centrifugation of venous blood (~700 rpm, 3 minutes). The upper plasma fraction rich in platelets and leukocytes was aspirated and applied to defect surfaces for approximately 5 minutes before flap closure.
  Other Names: Autologous Injectable PRF
  Arms: Test - OFD + EDTA + i-PRF

SUMMARY:
This study is designed to evaluate a new method to improve healing in patients with gum disease (periodontitis). A total of 42 adults with gum pockets deeper than 5 millimeters will take part. All patients will undergo flap surgery, which is a standard treatment for gum disease. Half of the patients will also receive an additional treatment with injectable platelet-rich fibrin (i-PRF), made from their own blood, together with root surface cleaning using EDTA gel. Patients will be followed for 6 months. The study will measure changes in gum pocket depth, gum attachment to teeth, and healing.

DETAILED DESCRIPTION:
Periodontitis is a chronic inflammatory disease of the tooth-supporting tissues. Open flap debridement (OFD) is a standard surgical approach for the management of deep periodontal pockets. Injectable platelet-rich fibrin (i-PRF) is an autologous, anticoagulant-free platelet concentrate prepared with low-speed centrifugation and characterized by a fibrin network that gradually releases growth factors. Neutral-pH 24% EDTA root-surface conditioning is used to remove the smear layer and expose collagen, which may support early cell attachment and the adsorption of bioactive molecules.

This single-center, randomized, parallel-group, open-label clinical trial is designed to evaluate whether the adjunctive use of i-PRF after EDTA root conditioning provides additional benefits compared with EDTA conditioning alone. Adults with periodontitis will be enrolled at a university periodontal clinic and randomized to one of two groups:

Control group: OFD with 24% EDTA gel conditioning (3 minutes)

Test group: OFD with 24% EDTA gel conditioning (3 minutes) followed by application of i-PRF retained on defect surfaces for 5 minutes

A mixed defect model (sites with both intrabony and horizontal components) will be included to reflect real-world clinical presentations.

All participants will receive standardized Phase I therapy before surgery. On the day of surgery, an antiseptic rinse will be performed, local anesthesia will be administered, full-thickness flaps will be elevated, and meticulous debridement/root planing will be completed. In the test arm, i-PRF will be prepared from venous blood collected into plain glass tubes and centrifuged at ~700 rpm (60 g) for 3 minutes; the platelet-rich upper layer (~1-1.5 mL per tube) will be aspirated and applied to the defect for 5 minutes before primary closure with 4-0 monofilament sutures. Postoperative care will include analgesic and/or anti-inflammatory medication as needed and an antiseptic mouthwash; systemic antibiotics will not be routinely prescribed. Sutures will be removed at approximately 1 week. A planned follow-up schedule will include weekly visits during the first month and monthly visits thereafter through month 6.

The primary outcome will be the change in probing pocket depth (PPD) at surgical sites at 6 months. Key secondary outcomes will include clinical attachment level (CAL), plaque and gingival indices, bleeding on probing, gingival recession depth and width, patient-reported pain and sensitivity (VAS), and postoperative clinical healing parameters such as edema, erythema, and necrosis, assessed at prespecified time points. Randomization will be computer-generated; surgeries and measurements will be performed by an experienced periodontist using calibrated probes.

The study has been approved by an institutional ethics committee and will be conducted in accordance with the Declaration of Helsinki and good clinical practice principles. The trial does not involve any U.S. FDA-regulated drug or device. An independent data monitoring committee will not be convened given the low-risk, single-center nature of the interventions; adverse events will be actively assessed at follow-up visits, and participants may withdraw at any time without penalty.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* Diagnosis of Stage II-IV periodontitis
* Presence of ≥3 adjacent teeth with probing pocket depth (PPD) ≥5 mm
* Systemically healthy individuals
* Non-smokers
* Ability and willingness to comply with oral hygiene instructions and study follow-up visits

Exclusion Criteria:

* Systemic diseases or conditions affecting periodontal healing (e.g., uncontrolled diabetes, immunodeficiency)
* Pregnancy or lactation
* Current or previous smokers
* Use of medications that may affect periodontal status (e.g., immunosuppressants, bisphosphonates)
* Previous periodontal treatment within the last 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Change in probing pocket depth (mm) at treated sites | Baseline and 6 months post-surgery
  Measured with a UNC-15 periodontal probe at treated sites.

SECONDARY OUTCOMES:
Change in clinical attachment level (mm) at treated sites | Baseline and 6 months post-surgery
  Measured with a UNC-15 periodontal probe.
Mean Plaque Index (Silness and Löe Index, 0-3 scale) | Baseline, 3 months, and 6 months
  Full-mouth plaque scores (0 = no plaque, 3 = abundant plaque). Higher scores indicate worse oral hygiene.
Mean Gingival Index (Löe and Silness Index, 0-3 scale) | Baseline, 3 months, and 6 months
  Gingival inflammation scores (0 = normal gingiva, 3 = severe inflammation). Higher scores indicate worse gingival condition.
Percentage of sites with bleeding on probing (%) | Baseline, 3 months, and 6 months
  Assessed by gentle probing (0 = no bleeding, 1 = bleeding present). Higher percentages indicate worse periodontal condition.
Change in gingival recession depth (mm) at treated sites | Baseline, 3 months, and 6 months
  Measured vertically from the cemento-enamel junction (CEJ) to the gingival margin using a periodontal probe.
Change in gingival recession width (mm) at treated sites | Baseline, 3 months, and 6 months
  Measured horizontally at the CEJ level using a periodontal probe.
Visual Analog Scale (VAS, 0-10) scores for pain and sensitivity | Immediately after surgery, Week 1, and Week 2
  Patient-reported outcomes (0 = no pain/sensitivity, 10 = worst imaginable). Higher scores indicate worse symptoms.
Clinical healing parameters (edema, erythema, necrosis) | Week 1, Week 2, and 1 month post-surgery
  Presence or absence assessed by clinical inspection.

CONTACTS AND LOCATIONS:
Overall Officials: HALİL A BIÇAKÇIOĞLU, PhD, Principal Investigator — Department of Periodontology, Faculty of Dentistry, Gazi University, Ankara, Turkey
Locations (1):
- Gazi University Faculty of Dentistry, Department of Periodontology, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to patient privacy considerations and institutional restrictions.